CLINICAL TRIAL: NCT00001839
Title: A Randomized Trial of Antithymocyte Globulin Versus Cyclosporine to Treat the Cytopenia of Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990021; 99-CC-0021
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1998-12

CONDITIONS: Hematologic Diseases; Myelodysplastic Syndromes
Keywords: Anemia; Immunosuppressive; Phase II Trial; Pre-Leukemia; Therapy; Myelodysplastic Syndrome
MeSH Terms: conditions — Hematologic Diseases; Myelodysplastic Syndromes; Anemia | interventions — Antilymphocyte Serum; Cyclosporine

INTERVENTIONS:
Drug: Antithymocyte globulin
Drug: Cyclosporine

SUMMARY:
Approximately 40% of the patients with myelodysplastic syndrome (MDS) die as a consequence of their cytopenia. As in aplastic anemia, the cytopenia of MDS may be partly due to cytotoxic T cell activity. Immunosuppressive therapy may therefore reverse the cytopenia. In a phase II pilot study of anti-thymocyte globin (ATG) to treat myelodysplastic syndrome (MDS); 41% of patients (61% of patients with refractory anemia) have responded in terms of transfusion independence. Recently, Jonasova et al [32] reported a 82% substantial hematological response rate in 18 patients with MDS of the refractory anemia (RA) subtype treated with cyclosporine alone. Just over 50% of the patients in this series had MDS of the hypocellular type. Cyclosporine alone if indeed efficacious would be a powerful therapeutic option that could be readily used by hematologists in the community to treat patients with MDS. This efficacy needs to be proven in a larger study which includes patients with the other subtypes of MDS and more patients with the non-hypocellular forms of MDS (which constitute approximately 70% of the cases in the community). As MDS is a heterogeneous group of disorders, a randomized comparison with the other immunomodulating intervention of proven benefit, ATG, is appropriate. In this randomized study patients with MDS will receive either ATG alone or cyclosporine alone.

DETAILED DESCRIPTION:
Approximately 40% of the patients with myelodysplastic syndrome (MDS) die as a consequence of their cytopenia. As in aplastic anemia, the cytopenia of MDS may be partly due to cytotoxic T cell activity. Immunosuppressive therapy may therefore reverse the cytopenia. In a phase II pilot study of anti-thymocyte globulin (ATG) to treat myelodysplastic syndrome (MDS); 41% of patients (61% of patients with refractory anemia) have responded in terms of transfusion independence. Recently, Jonasova et al [32] reported a 82% substantial hematological response rate in 18 patients with MDS of the refractory anemia (RA) subtype treated with cyclosporine alone. Just over 50% of the patients in this series had MDS of the hypocellular type. Cyclosporine alone if indeed efficacious would be a powerful therapeutic option that could be readily used by hematologists in the community to treat patients with MDS. This efficacy needs to be proven in a larger study which includes patients with the other subtypes of MDS and more patients with the non-hypocellular forms of MDS (which constitute approximately 70% of the cases in the community). As MDS is a heterogeneous group of disorders, a randomized comparison with the other immunomodulating intervention of proven benefit, ATG, is appropriate. In this randomized study patients with MDS will receive either ATG alone or cyclosporine alone.

ELIGIBILITY:
MDS of RA & RAEB sub-types.

No current treatment and off other treatments for at least two weeks.

ECOG performance status less than or equal to 2.

No MDS of FAB sub-group' refractory anemia with ring sideroblasts' (RARS).

No transforming to acute leukemia (FAB sub-group RAEB-Tie.; greater than 20% blasts in marrow aspirate).

No hypoplastic marrow without one major or two minor criteria as outlined in table 3 of the appendix.

No one being treatment with growth factors or cyclosporine within four weeks prior to entry to protocol.

No previous treatment with ATG.

No ECOG performance status of greater than 2.

No active uncontrolled infection.

No women which current pregnancy, or unwilling to take oral contraceptives if of childbearing potential.

No patients for whom bone marrow transplant is indicated as primary therapy.

No one age less than 18 years.

Must be able to give informed consent.

No HIV positive patients.

No active malignant disease (excluding basal cell carcinoma).

No one with serum creatine greater than 2mg/dl.

No patients who are moribund or patients with concurrent hepatic, renal, cardiac, metabolic, or any disease of such severity that death within 7-10 days is likely.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182
Dates: Start 1998-12; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States